CLINICAL TRIAL: NCT02739126
Title: Comparing the Diagnostic Yield of Radial Endo-Bronchial Ultra-Sound Guided Biopsy When Using a Thick (1.7mm) With an Aspiration Needle Biopsy Vs. a Thin USS Probe (1.4mm), in Peripheral Lung Lesions.
Brief Title: Comparing the Diagnostic Yield of Radial EBUS Guided Biopsies When Using a Thick (1.7mm) Vs. Thin (1.4 mm) USS Probe.
Acronym: R-EBUST2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Middlemore Hospital, New Zealand (Other)
Responsible Party: Principal Investigator, Samantha Herath, Respiratory Physician, Middlemore Hospital, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: R- EBUST 2
Record Dates: First submitted 2016-02-19; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Pulmonary Parenchymal Lesions
Keywords: Diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thick USS (1.7mm) with use of additional aspiration needle (Active Comparator)
  Interventions: Procedure: Radial EBUS biopsy; Device: Types of Radial Ultrasound probes
- Thin USS (1.4mm) (Active Comparator)
  Interventions: Procedure: Radial EBUS biopsy; Device: Types of Radial Ultrasound probes

INTERVENTIONS:
Procedure: Radial EBUS biopsy — Radial EBUS is an endobronchial USS which is used to obtain biopsies from a peripheral lung mass.
Device: Types of Radial Ultrasound probes — The Radial USS probe comes in two sizes. A thick USS probe that is 1.7mm and the thin USS is 1.4mm in diameter.

SUMMARY:
Obtaining a tissue sample to diagnose parenchymal lung lesions (PPL) suspected of cancerous origin is of utmost importance. Due to it's markedly favourable safety profile, a bronchoscopic biopsy method called Radial EBUS is becoming increasingly popular. However, a meta-analysis reports the success rate of Radial EBUS in diagnosis is 73%, which in comparison to CT guided biopsy which is the gold standard in diagnosing PPL (90% success rate), is sub-optimal.

There are 2 types of USS probes used in the R-EBUS procedure. Whilst the thicker USS probe (1.7mm) is capable of accommodating larger biopsy instruments, the thinner USS probe could be advanced more peripherally to obtain a biopsy.

Therefore identifying what type of USS probe is better for a given PPL will aid in improving the diagnostic yield.

In this study, investigators compare these two types of probes in the ability to diagnose a PPL.

The biopsy instruments used for both arms are forceps and cytology brush. For the thick USS arm, in addition, an aspiration needle will also be used. (The thin USS guide sheath is too small to accommodate an aspiration needle)

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for R-EBUS as per routine management.
* Patient judged to be medically stable to give consent for this study.

Exclusion Criteria:-Unsuitable for flexible bronchoscopy and biopsy

* INR>1.5
* Platelets<150.
* Hb> 80g/l
* Liver function tests (AST/ALT) <2 times upper limit of normal
* Neutrophil count >1.0
* EGFR >30ml/kg/min
* On anticoagulation, that cannot be withheld for the procedure, due to medical reasons (e.g. On-clopidogrel with recent drug-eluting stent placement.)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Comparing the diagnostic yield (sensitivity) from the biopsies taken using the thick USS and Guide sheath to that of biopsies taken using the thin USS and Guide sheath. | 18 months
  A blinded pathologist will assess all samples from the thick USS arm and all samples from the thin USS arm separately and come to a conclusion as
  1. To what biopsies give a diagnosis of malignancy and
  2. Will decide what is the best sample in comparing all samples from both arms defined as " the highest number of malignant cells/hpf".

SECONDARY OUTCOMES:
Suitability of the biopsy samples from each arm to perform EGFR mutation testing. | 18 months
  A blinded pathologist will assess all samples from the thick USS arm and all samples from the thin USS arm separately and come to a conclusion as to what is the best sample defined as " the sample most suitable for EGFR mutation analysis".
Compare the procedure related bleeding and pneumothorax rates between the two arms. | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Middlemore Hospital, Counties Manakau District Health Board, Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No